CLINICAL TRIAL: NCT03154424
Title: Bridging Versus Non-bridging Dynamic External Fixation in Early Total Care Treatment Unstable Distal Radius Fractures in Elderly Polytrauma Patients: A Randomized Controlled Study
Brief Title: Dynamic External Fixation in Treatment Distal Radius Fractures - Elderly Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Faculdade de Medicina do ABC (Other)
Responsible Party: Principal Investigator, Marcio Aurelio Aita, Affiliated Professor, Faculdade de Medicina do ABC
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 32925713.9.0000.0082
Record Dates: First submitted 2017-05-11; First posted 2017-05-16 (Actual); Last update posted 2017-05-16 (Actual); Status verified 2017-05

CONDITIONS: Distal Radius Fracture; Multiple Trauma; Elderly Person Maltreatment
MeSH Terms: conditions — Wrist Fractures; Multiple Trauma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Patients were randomized by drawing lots currency (Face = A - treatment with fixation "non-bridging"; Crown = B - Treatment with the method "bridging"), which were printed and placed in sealed envelopes before the study started.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bridging (control group) (Placebo Comparator): External fixation in treatment the distal radius fracture
  Interventions: Procedure: External fixation in treatment the distal radius fracture
- Nonbridging (tested group) (Active Comparator): External fixation in treatment the distal radius fracture improve grip strength?
  Interventions: Procedure: External fixation in treatment the distal radius fracture

INTERVENTIONS:
Procedure: External fixation in treatment the distal radius fracture — Compare two techniques

SUMMARY:
A single center, parallel group, prospective, randomized clinical trial was conducted at the department of Hand Surgery, ABC (Andre, Bernardo, Caetano) Foundation University Hospital, Santo Andre, Brazil. Two implants used for fixation in closed reduction of distal radius fractures were compared: the bridging dynamic Galaxy Wrist external fixator (Orthofix®, Verona) and the non-bridging Galaxy wrist external fixator system (Orthofix®, Verona).

DETAILED DESCRIPTION:
Dynamic external fixator in the ETC (Early Total Care) of unstable DRFs (distal radius fractures) may be a good choice of treatment. Because it's fast, safe, minimally invasive and easily performed method, it could help in the inflammatory systemic response to trauma, unable earlier functional recovery and shorten the hospitalization time of these patients (elderly and polytrauma). From this, in this study to obtain relevant information about each type of treatment, avoid possible selection bias, information and confusion. Choose a reproducible and effective method (external fixator), which presents a cost / benefit compatible with our reality, but that generates doubt the best way to apply this "bridging" which is already used and that will be our control group and "non-bridging", which will be the group to be tested.

Rather than establishing the actual value of each of these procedures, is necessary to optimize and improve the quality of life of these patients in order to return to your personal and professional activities as soon as possible.

ELIGIBILITY:
Inclusion Criteria:

* skeletally mature patients, elderly (60 y.o. or more)
* all with a diagnosis of unstable distal radius fractures (AO type A or C)
* associated a multiple injured ( polytrauma ).

Exclusion Criteria:

* ongoing chemo or radiotherapy,
* mental illness,
* alcohol abuse.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2017-05-01 (Actual); Study Completion 2017-05-01 (Actual)

PRIMARY OUTCOMES:
Grip strenght | 12 months
  use the specific Jamar Hand Dynamometer to measure the arc of movement the wrist

SECONDARY OUTCOMES:
range of wrist motion | 12 months
  use the specific goniometer to measure the arc of movement the wrist
Radiograph assesment | 12 months
  Measure ulna and radial shortening, tilt palmar
DASH Questionnaire | 12 months
  measure life quality
VAS (visual analog scale) | 12 months
  patient reported outcome (pain) in scale interval (0 until 10)

IPD SHARING:
Plan to Share IPD: No